CLINICAL TRIAL: NCT06571188
Title: Comparison of Ultrasound-Guided Continuous Erector Spinae Plane Block Versus Thoracic Epidural Analgesia in Postoperative Analgesia Following Thoracotomy Surgeries: a Randomised Trial
Brief Title: Comparison of Ultrasound-Guided Continuous Erector Spinae Plane Block Versus Thoracic Epidural Analgesia
Acronym: TEAVSESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 8/2024ANET6-1
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-08

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups according to the 1:1 ratio of ESPB group and TEB group. A research coordinator is designated to distribute and preserve randomization result. The coordinator will open the envelopes for allocation according to the order of enrolment and prepare the study drug
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The random sequence will be sealed in consecutively numbered opaque envelopes and kept by the study coordinator.
  Participants will be randomly divided into two groups . The coordinator will open the envelopes for allocation according to the order of enrolment and prepare the study drug.
  The participants will be blinded to the allocation.Anaesthesiologists who perform the nerve block and take charge of intraoperative management and surgeons are independent individuals.Researchers who do not take part in the nerve block and intraoperative management are designated to postoperative follow-up. Besides, trained anaesthesiologist who do not perform the block will be designated to evaluate the clinical features of the block objectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEB GROUP (Active Comparator): In group TEB, The epidural catheter will be inserted preoperatively at the T5-T7 vertebral level; the exact level will be at the discretion of the attending anaesthesiologist. A loading dose of bupivacaine 0.25% (max 10 ml) will be administered, followed by an intraoperative infusion of bupivacaine 0.125 % with Fentanyl 1 μg/ml.].
  Interventions: Other: THORACIC EPIDURAL BLOCK
- ESPB group (Active Comparator): In group ESPB, The ESP block will be performed as described by Forero et al. A Tuohy needle will be inserted with an in-plane technique in a caudal to cephalad direction until bony contact with the transverse process is obtained. Hydro dissection with normal saline will be performed to identify and open up the correct plane for injection. A loading dose of Bupivacaine will be injected followed by the insertion of an 18-g catheter 5 cm beyond the needle tip. No further local anaesthetic will be administered intra-operatively. Following the end of surgery, a continuous infusion of 5 ml/h of Bupivacaine 0.125%, supplemented by a 10-ml bolus injection every 3 h, will be administered through the ESPB catheter
  Interventions: Other: ERECTOER SPINE BLOCK

INTERVENTIONS:
Other: THORACIC EPIDURAL BLOCK — In group TEB, The epidural catheter will be inserted preoperatively at the T5-T7 vertebral level; the exact level will be at the discretion of the attending anaesthesiologist. A loading dose of bupivacaine 0.25% (max 10 ml) will be administered, followed by an intraoperative infusion of bupivacaine 0.125 % with fentanyl 1 μg/ml.].
  Other Names: TEB
  Arms: TEB GROUP
Other: ERECTOER SPINE BLOCK — The ESP block will be performed as described by Forero et al
  Other Names: ESPB
  Arms: ESPB group

SUMMARY:
There are limited studies comparing these two modalities ( thoracic epidural and erector spine block) for relieving the pain after thoracic surgeries .this study aim to investigate this purpose

DETAILED DESCRIPTION:
The random sequence will be sealed in consecutively numbered opaque envelopes and kept by the study coordinator. Participants will be randomly divided into two groups according to the 1:1 ratio of ESPB group and TEB group. A research coordinator is designated to distribute and preserve randomization result. The coordinator will open the envelopes for allocation according to the order of enrolment and prepare the study drug.

The participants will be blinded to the allocation. Because the needle injection of ESPB and TEB are very close, participants themselves could hardly detect the clinical differences. Anaesthesiologists who perform the nerve block and take charge of intraoperative management and surgeons are independent individuals. Only the random sequence number rather than the specific nerve block type will be recorded in the electronic anaesthesia information management system .Researchers who do not take part in the nerve block and intraoperative management are designated to postoperative follow-up. Besides, trained anaesthesiologist who do not perform the block will be designated to evaluate the clinical features of the block objectively

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be from18-70 years old with ( American association of anaesthesiologist) ASA physical status I to III scheduled for elective thoracic surgeries.

Exclusion Criteria:

* Patients who are:
* Unable to cooperate.
* Patients who have allergy to any of the study drugs.
* Patients who are on opioids.
* Local infection at the site of injection or systemic infection.
* Patients with coagulation disorders or on anticoagulation therapy Unable to communicate preoperatively due to severe dementia, language barrier, or neuropsychiatric disorder
* Unable to perform nerve block procedure due to difficult anatomy through ultrasound scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
MORPHINE CONSUMPTION | 24 hours
  cumulative 24 h opioid (morphine) consumption
Numeric rating scale | 24 hours
  is an 11-point scale scored from 0-10:
  1. "0" = no pain
  2. "10" = the most intense pain imaginable Patients verbally select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours.

SECONDARY OUTCOMES:
Time for first rescue analgesia | 24 hours
  Time for first rescue analgesia will be measured and recorded
The number of rescue analgesics | 24 hours
  the number of rescue analgesics within 24hrs after surgery will be recorded
Time to ambulation | 24 hours
  Time to ambulation WILL BE RECOREDED
Complications | 24 hours
  Complications like bradycardia or hypotension, itching, nausea and vomiting will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No